CLINICAL TRIAL: NCT07252362
Title: LCMS-Based Metabolic Analysis Explores the Effect of American Ginseng on Urine and Plasma in Healthy Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, baoguanai, attending doctor, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021KY577
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: The Impact of American Ginseng on the Metabolomics of Urine and Plasma in Healthy Individuals
Keywords: American ginseng; metabolomics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- American Ginseng group (Other): All the subjects took 3 grams of American ginseng half an hour after breakfast every day for 14 consecutive days.
  Interventions: Other: American Gginseng

INTERVENTIONS:
Other: American Gginseng — All the subjects took 3 grams of ginseng half an hour after breakfast every day for 14 consecutive days.

SUMMARY:
Researchers will use LCMS Metabolic Analysis to Explore the Effect of American Ginseng on Urine and Plasma in Healthy Individuals

Participants will:

* Take 3 grams of American Ginseng powder every day for 14 days
* Collect the fasting urine samples at the following times at the hospital: On the first day, on the 7th day after taking the medicine, and on the 14th day after taking the medicine.
* Collect the fasting Serum samples at the following times at the hospital: On the first day and on the 14th day after taking the medicine.
* Have their any adverse effects monitored and evaluated throughout the study.

ELIGIBILITY:
* 18 to 45 years old;

  * The subjects were fully informed about the research process and signed the informed consent form (the subjects had no abnormalities in routine physical examinations, no previous medical history, and no history of drug allergies); ③ During the trial, they were required to have a light diet and were prohibited from consuming alcoholic and caffeinated beverages;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Urine metabolomics | From enrollment to the end of treatment at 2 weeks
  By using LCMS Metabolic Analysis to Explore the Effect of American Ginseng on Urine in Healthy Individuals

SECONDARY OUTCOMES:
Plasma metabolomics | From enrollment to the end of treatment at 2 weeks
  By using LCMS Metabolic Analysis to Explore the Effect of American Ginseng on plasma in Healthy Individuals.

CONTACTS AND LOCATIONS:
Overall Officials: guan ai Bao, Master, Study Director — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No